CLINICAL TRIAL: NCT07363083
Title: Predictors of Treatment Response to Greater Occipital Nerve Pulsed Radiofrequency in Older Patients With Chronic Migraine
Brief Title: Treatment Response to GON Pulsed Radiofrequency in Elderly Patients With Chronic Migraine
Acronym: FRAIL-GON
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Assoc. Prof., Ankara City Hospital Bilkent
Other Study IDs: 111213
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Headache, Migraine
Keywords: Migraine Headache; Elderly, Frail; Nerve Blockade
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GON_PRF group: This study is a single-center, prospective, single-arm interventional clinical trial designed to evaluate the effectiveness of greater occipital nerve pulsed radiofrequency (GON-PRF) treatment and to identify predictors of treatment response in patients aged 65 years and older with a diagnosis of chronic migraine. Within the scope of the study, patients presenting to the algology clinic who meet the inclusion criteria will undergo ultrasound-guided GON-PRF treatment in accordance with standard clinical practice.

SUMMARY:
Headache disorders are highly prevalent in older adults, yet their management remains challenging due to comorbidities, polypharmacy, and the paucity of evidence derived from geriatric populations. Most randomized clinical trials exclude elderly patients, underscoring the need for effective and safe non-pharmacological treatment strategies for headache in this age group.

Greater occipital nerve blocks are commonly used in the treatment of migraine and other headache disorders; however, their clinical benefit is often transient. Pulsed radiofrequency (PRF) has been introduced as a minimally invasive technique aimed at prolonging therapeutic effects through neuromodulation without causing structural neural damage. Although greater occipital nerve pulsed radiofrequency (GON-PRF) has demonstrated efficacy in various headache disorders, its effectiveness in patients aged 65 years and older has not been adequately investigated.

The primary aim of this study is to evaluate the effectiveness of GON-PRF in patients aged ≥65 years with chronic migraine by assessing changes in pain intensity, monthly headache days, and monthly severe headache days. The secondary aim is to identify geriatric predictors of treatment response, including frailty status and the Geriatric Nutritional Risk Index (GNRI), in order to support individualized treatment strategies for older adults.

DETAILED DESCRIPTION:
Headache disorders are common across all age groups. As the global population ages, the number of older adults affected by headache disorders continues to rise, and an increasing proportion of elderly individuals seek medical care for headache-related complaints. Although primary headache disorders remain prevalent in this population, secondary causes must always be excluded as a first step. Previous estimates suggest that the one-year prevalence of primary headache disorders in adults aged 55-94 years is approximately 40.5% (1).

The management of headache in geriatric patients is often complex and challenging, requiring careful consideration of multiple factors, including comorbidities, polypharmacy, potential drug interactions, and age-related adverse effects. Moreover, evidence guiding headache treatment in older adults is limited, as most published clinical trials have excluded elderly populations. Consequently, there is a clear need for effective treatment options for headache in older adults, particularly non-pharmacological approaches that are less influenced by comorbid conditions and medication burden.

Peripheral nerve blocks, particularly greater occipital nerve blocks (GONB), have long been used in the treatment of various headache disorders and cranial neuralgias, including migraine, cluster headache, and cervicogenic headache, and may represent a safe alternative to standard pharmacotherapy in this demographic. In a retrospective study by Hascalovici et al., which evaluated the demographic, clinical, and therapeutic characteristics of patients aged 65 years and older treated with peripheral nerve blocks (greater and/or lesser occipital, auriculotemporal, supraorbital, and supratrochlear nerves), peripheral nerve blocks were reported to be a safe and effective headache management strategy for older adults (2).

Although greater occipital nerve blocks performed with local anesthetics and/or corticosteroids have demonstrated clinical benefit in the treatment of headache disorders, the duration of their efficacy is often limited. Pulsed radiofrequency (PRF) therapy has been introduced as a minimally invasive technique to prolong therapeutic effects. PRF modulates pain transmission by generating an electric field at the targeted nerve without causing structural damage to neural tissue or surrounding structures (3). A recent systematic review evaluating the efficacy and safety of greater occipital nerve pulsed radiofrequency in headache disorders reported that GON-PRF was effective in reducing pain intensity and headache frequency across various primary headache conditions, with a favorable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older

Diagnosis of chronic migraine according to ICHD criteria

Presentation to the algology clinic

Eligibility for greater occipital nerve pulsed radiofrequency (GON-PRF) treatment according to the study protocol

Ability to provide written informed consent

Exclusion Criteria:

* Acute headache or pain conditions

Malignancy-related headache

Severe cognitive or communication impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65 years or over patients with chronical migraine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | baseline, 1st month, 3rd month
  VAS: Pain intensity, assessed by the Visual Analog Scale
Primary outcme | baseline, 1st month, 3rd month
  Monthly headache frequency
Primary outcome | baseline, 1st month, 3rd month.
  Number of headache days per month

SECONDARY OUTCOMES:
secondary outcome | baseline
  Baseline frailty index
secondary outcome | baseline
  Baseline nutritional index (GNRI)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park D, Chang MC. The mechanism of action of pulsed radiofrequency in reducing pain: a narrative review. J Yeungnam Med Sci. 2022 Jul;39(3):200-205. doi: 10.12701/jyms.2022.00101. Epub 2022 Apr 7. PMID 35385898